CLINICAL TRIAL: NCT00002597
Title: A PHASE III TRIAL OF THE STUDY OF ENDOCRINE THERAPY USED AS A CYTOREDUCTIVE AND CYTOSTATIC AGENT PRIOR TO RADIATION THERAPY IN GOOD PROGNOSIS LOCALLY CONFINED ADENOCARCINOMA OF THE PROSTATE
Brief Title: Radiation Therapy With or Without Antiandrogen Therapy in Treating Patients With Stage I or Stage II Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-9408; CDR0000063821
Record Dates: First submitted 1999-11-01; First posted 2004-02-27 (Estimated); Results first posted 2017-06-06 (Actual); Last update posted 2018-06-14 (Actual); Status verified 2018-05

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Flutamide; Goserelin; Leuprolide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Neoadjuvant TAS + RT (Experimental): Neoadjuvant total androgen suppression (TAS) - Flutamide and Zoladex or Lupron - two months before and during radiation therapy.
  Interventions: Drug: flutamide; Drug: Zoladex; Drug: Lupron; Radiation: radiation therapy
- Radiation therapy alone (Other): Radiation therapy alone
  Interventions: Radiation: radiation therapy

INTERVENTIONS:
Drug: flutamide — Two 125 mg capsules (t.i.d., p.o.) beginning two months before RT and continuing until RT is completed.
  Other Names: Eulexin
  Arms: Neoadjuvant TAS + RT
Drug: Zoladex — 3.6 mg s.c. monthly x 4 beginning two months before RT and continuing until RT is completed. The 3-month preparation may be used instead of three separate monthly injections.
  Other Names: goserelin acetate
  Arms: Neoadjuvant TAS + RT
Drug: Lupron — 7.5 mg IM (intramuscular) monthly x 4 beginning two months before RT and continuing until RT is completed. The 3-month preparation may be used instead of three separate monthly injections.
  Other Names: leuprolide acetate
  Arms: Neoadjuvant TAS + RT
Radiation: radiation therapy — 46.8 Gy (1.8 Gy/day four to five times a week [26 fx]) to regional lymphatics followed by 19.8 Gy (1.8 Gy/day x 11 fx) for a total of 66.6 Gy to the prostate. Prostate only may be treated in defined circumstances.

SUMMARY:
RATIONALE: Radiation therapy (RT) uses high-energy x-rays to damage tumor cells. Androgens can stimulate the growth of prostate cancer cells. Hormone therapy using flutamide, goserelin, and leuprolide may fight prostate cancer by reducing the production of androgens. It is not yet known which regimen of antiandrogen therapy is most effective for prostate cancer.

PURPOSE: Randomized phase III trial to study the effectiveness of radiation therapy with or without antiandrogen therapy in treating patients who have stage I or stage II prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES: Primary: To evaluate whether a combination of Zoladex and flutamide used as cytoreductive agents prior to and during definitive radiation therapy improves overall survival over radiation therapy alone in locally confined carcinomas of the prostate; Secondary: To compare the rates of disease-specific survival, clinical relapse (local progression and/or distant failure), freedom from prostate-specific antigen (PSA) failure, freedom from second clinical relapse, freedom from second PSA relapse, and disease-free survival; To compare the prostate re-biopsy at two years; To measure the effect on sexual function.

OUTLINE: This is a randomized, multicenter study. Patients were stratified by PSA level (less than 4 vs 4-20), tumor differentiation (well vs moderate vs poor), nodal status (N0 [nodes evaluated by surgical sampling] vs NX [nodes evaluated negative by imaging methods only]), and participating center. Patients are randomized to one of two treatment arms. Arm I: Patients receive oral flutamide 3 times a day and goserelin subcutaneously once every 4 weeks, or once as a time release injection (intramuscular leuprolide may be substituted for goserelin), beginning 2 months prior to radiotherapy and continuing until completion of radiotherapy. Patients undergo radiotherapy daily 4-5 days per week for almost 8 weeks. Arm II: Patients undergo radiotherapy only, as in arm I. Patients are followed every 3 months for the remainder of the first year, every 4 months for the second year, every 6 months for the third through fifth years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 1980 patients within 5 years.

ELIGIBILITY:
Inclusion criteria:

* Histologically confirmed locally confined adenocarcinoma of the prostate with primary tumors confined to the prostate, clinical stage T1b,1c, 2a or 2b.
* Negative nodes evaluated by imaging methods (classified in the study as NX) or by surgical sampling (classified in the study as N0).
* Karnofsky performance status ≥ 70.
* PSA is mandatory, must be ≤ 20)
* No prior hormonal therapy, radiation or chemotherapy.
* Prior finasteride for prostate hypertrophy allowed if discontinued at least 60 days prior to randomization.
* Prior testosterone administration allowed if at least 90 days elapsed since last administration.
* No evidence of distant metastasis or other synchronous primary. Patients with prior invasive malignancy who were disease free for at least 5 years could be eligible with pre-randomization approval by the study chairman.
* Treatment begins within 21 days after randomization.
* Patients signs a study-specific informed consent form.
* Alanine Aminotransferase (ALT) within 2x upper normal limits.

Exclusion criteria:

* Stage T1a or ≥ T2c disease.
* Lymph node involvement (N1 - N3).
* Evidence of distant metastasis. (M1)
* PSA > 20.
* Radical surgery or cryosurgery for carcinoma of the prostate, previous irradiation, antiandrogen therapy or chemotherapy.
* Previous or concurrent cancers other than basal cell or squamous cell skin carcinoma.

Patients with squamous cell carcinomas required to be NED (no evidence of disease) for a minimum of two years prior to study entry.

* Major medical or psychiatric illness which, in the investigator's opinion, would prevent completion of treatment and would interfere with follow-up.
* Karnofsky performance status of < 70.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2028 (Actual)
Dates: Start 1994-10; Primary Completion 2011-07 (Actual); Study Completion 2018-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David G. McGowan, MD, Study Chair — Cross Cancer Institute at University of Alberta
Locations (239):
- United States (222):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Huntsville Hospital System, Huntsville, Alabama
  - Comprehensive Cancer Institute of Huntsville, Huntsville, Alabama
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - Alabama Oncology, LLC, Montgomery, Alabama
  - Radiation Oncology Associates of West Alabama, Tuscaloosa, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Arizona Cancer Center, Tucson, Arizona
  - Mount Diablo Medical Center, Concord, California
  - Cancer Center and Beckman Research Institute, City of Hope, Duarte, California
  - California Cancer Center, Fresno, California
  - Saint Agnes Cancer Center, Fresno, California
  - Glendale Memorial Hospital and Health Center, Glendale, California
  - Sutter Health Western Division Cancer Research Group, Greenbrae, California
  - University of California San Diego Cancer Center, La Jolla, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Veterans Affairs Medical Center - Long Beach, Long Beach, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Cancer Care Center, Pomona, California
  - Radiation Oncology Center - Sacramento, Sacramento, California
  - Radiation Medical Group, Inc., San Diego, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - O'Connor Hospital, San Jose, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - Memorial Hospital Cancer Center, Colorado Springs, Colorado
  - University of Colorado Cancer Center, Denver, Colorado
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Lykes Center for Radiation Therapy, Clearwater, Florida
  - Halifax Medical Center, Daytona Beach, Florida
  - Radiation Therapy Associates - Fort Myers, Fort Myers, Florida
  - University of Florida Health Science Center, Gainesville, Florida
  - Health First Holmes Regional Medical Center, Melbourne, Florida
  - dVeterans Affairs Medical Center - Miami, Miami, Florida
  - Sylvester Cancer Center, University of Miami, Miami, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Radiation Oncology Group, Orange Park, Florida
  - MD Anderson Cancer Center Orlando, Orlando, Florida
  - Bay Medical Center, Panama City, Florida
  - Gulf Coast Cancer Treatment Center, Panama City, Florida
  - Sarasota Radiation and Medical Oncology Center, Sarasota, Florida
  - Tallahassee Memorial Healthcare, Tallahassee, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Medical Center/John B. Amos Community Cancer Center, Columbus, Georgia
  - InterCommunity Cancer Center at Rome, Rome, Georgia
  - Northwest Community Hospital, Arlington Heights, Illinois
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - Provena St. Joseph Hospital- Regional Cancer Care Center, Elgin, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - St. John's Medical Center, Anderson, Indiana
  - Veterans Affairs Medical Center - Indianapolis (Roudebush), Indianapolis, Indiana
  - Clarion Health Partners Inc., Indianapolis, Indiana
  - Community Hospitals of Indianapolis - Regional Cancer Center, Indianapolis, Indiana
  - Ball Memorial Hospital, Muncie, Indiana
  - Wendt Regional Cancer Center of Finley Hospital, Dubuque, Iowa
  - Holden Comprehensive Cancer Center at The University of Iowa, Iowa City, Iowa
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - Louisville Radiation Oncology, Louisville, Kentucky
  - Merle M. Mahr Cancer Center, Madisonville, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Romagosa Radiation Oncology Center, Lafayette, Louisiana
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Maine Medical Center, Portland, Maine
  - Anne Arundel Oncology Center, Annapolis, Maryland
  - Greater Baltimore Medical Center and Cancer Center, Baltimore, Maryland
  - Harbor Hospital Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - Radiation Oncology Affiliates of Maryland, P.A., Baltimore, Maryland
  - Peninsula Regional Medical Center, Salisbury, Maryland
  - Cape Cod Hospital, Hyannis, Massachusetts
  - Veterans Affairs Medical Center - Boston (Jamaica Plain), Jamaica Plain, Massachusetts
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - McLaren Regional Cancer Center, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - Marquette General Hospital, Marquette, Michigan
  - MidMichigan Medical Center - Midland, Midland, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - St. Mary's Medical Center, Saginaw, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - North Mississippi Medical Center/Cancer Center, Tupelo, Mississippi
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Cancer Research for the Ozarks, Springfield, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - Mallinckrodt Institute of Radiology, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Nebraska Health System, Omaha, Nebraska
  - Methodist Cancer Center - Omaha, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Elliot Regional Cancer Center, Manchester, New Hampshire
  - Cooper Cancer Institute, Camden, New Jersey
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - John F. Kennedy Medical Center, Edison, New Jersey
  - Trinitas Hospital - Jersey Street Campus, Elizabeth, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - South Jersey Regional Cancer Center, Millville, New Jersey
  - Fox Chase Cancer Center at Virtua Memorial Hospital Burlington County, Mount Holly, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Atlantic City Medical Center, Pomona, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - Capital Health System at Mercer, Trenton, New Jersey
  - St. Francis Medical Center, Trenton, New Jersey
  - Associated Radiologists, P.A., Warren Township, New Jersey
  - Saint Joseph Medical Center, Albuquerque, New Mexico
  - Cancer Center of Albany Medical Center, Albany, New York
  - State University of New York Health Science Center at Brooklyn, Brooklyn, New York
  - New York Methodist Hospital, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Finger Lakes Radiation Oncology, P.C., Clifton Springs, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Beth Israel Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Champlain Valley Physicians Hospital Medical Center, Plattsburgh, New York
  - Vassar Brothers Hospital, Poughkeepsie, New York
  - University of Rochester Cancer Center, Rochester, New York
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Northeast Medical Center, Concord, North Carolina
  - East Carolina University School of Medicine, Greenville, North Carolina
  - Catawba Memorial Hospital, Hickory, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Meritcare Roger Maris Cancer Center, Fargo, North Dakota
  - Akron General Medical Center, Akron, Ohio
  - Akron City Hospital, Akron, Ohio
  - Christ Hospital, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - St. Anthony Hospital, Oklahoma City, Oklahoma
  - St. John Health System, Tulsa, Oklahoma
  - CCOP - Columbia River Program, Portland, Oregon
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - St. Luke's Hospital Regional Cancer Center, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Mercy Catholic Medical Center, Mercy Fitzgerald Divison, Darby, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Penn State Geisinger Cancer Center, Hershey, Pennsylvania
  - Hahnemann University Hospital, Philadelphia, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Veterans Affairs Medical Center - Philadelphia, Philadelphia, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Mercy Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Reading Hospital and Medical Center, Reading, Pennsylvania
  - Mercy Hospital Cancer Center - Scranton, Scranton, Pennsylvania
  - Wilkes Barre General Hospital, Wilkes-Barre, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - York Hospital, York, Pennsylvania
  - Roger Williams Medical Center/BUSM, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Jackson-Madison County General Hospital, Jackson, Tennessee
  - University of Tennessee, Memphis Cancer Center, Memphis, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Harrington Cancer Center, Amarillo, Texas
  - Julie and Ben Rogers Cancer Institute, Beaumont, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Wilford Hall - 59th Medical Wing, Lackland Air Force Base, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - Bayshore Medical Center, Pasadena, Texas
  - East Texas Medical Center - Cancer Institute, Tyler, Texas
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center, St. George, Utah
  - CCOP - Southwestern Vermont Regional Cancer Center, Bennington, Vermont
  - Vermont Cancer Center, Burlington, Vermont
  - Green Mountain Oncology Group, Rutland, Vermont
  - Martha Jefferson Hospital, Charlottesville, Virginia
  - Cancer Center at the University of Virginia, Charlottesville, Virginia
  - RMH Regional Canter Center, Harrisonburg, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Deaconess Medical Center, Spokane, Washington
  - Yakima Valley Memorial Hospital, Yakima, Washington
  - Schiffler Cancer Center, Wheeling, West Virginia
  - St. Vincent Hospital, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Foundation, La Crosse, Wisconsin
  - Southern Wisconsin Radiotherapy Center, Madison, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Community Memorial Hospital, Menomonee Falls, Wisconsin
  - St. Joseph's Hospital, Milwaukee, Wisconsin
  - Columbia Hospital, Milwaukee, Wisconsin
  - St. Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee (Zablocki), Milwaukee, Wisconsin
  - Southeastern Wisconsin Regional Cancer Center, Racine, Wisconsin
  - Waukesha Memorial Hospital, Waukesha, Wisconsin
- Canada (17):
  - Tom Baker Cancer Center - Calgary, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Newfoundland Cancer Treatment and Research Foundation, St. John's, Newfoundland and Labrador
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Northeastern Ontario Regional Cancer Centre, Sudbury, Greater Sudbury, Ontario
  - Cancer Care Ontario-Hamilton Regional Cancer Centre, Hamilton, Ontario
  - Kingston Regional Cancer Centre, Kingston, Ontario
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Ottawa Regional Cancer Centre - General Campus, Ottawa, Ontario
  - Northwestern Ontario Regional Cancer Centre, Thunder Bay, Thunder Bay, Ontario
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - CHUS-Hopital Fleurimont, Fleurimont, Quebec
  - McGill University, Montreal, Quebec
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

REFERENCES:
- [Background] Bruner D, Scott C, McGowan D, et al.: Factors influencing sexual outcomes in prostate cancer patients enrolled on radiation therapy oncology group studies 90-20 and 94-08. [Abstract] Proceedings of the International Society for Quality of Life Research 7: 575, 1998.
- [Background] Bruner DW, Scott CB, McGowan D, et al.: Validation of the sexual adjustment questionnaire (SAQ) in prostate cancer patients enrolled on Radiation Therapy Oncology Group studies 90-20 and 94-08. [Abstract] Int J Radiat Oncol Biol Phys 42 (suppl 1): A-156, 202, 1998.
- [Background] Johnke RM, Edwards JM, Evans MJ, Nangami GN, Bakken NT, Kilburn JM, Lee TK, Allison RR, Karlsson UL, Arastu HH. Circulating cytokine levels in prostate cancer patients undergoing radiation therapy: influence of neoadjuvant total androgen suppression. In Vivo. 2009 Sep-Oct;23(5):827-33. PMID 19779119
- [Result] Jones CU, Hunt D, McGowan DG, Amin MB, Chetner MP, Bruner DW, Leibenhaut MH, Husain SM, Rotman M, Souhami L, Sandler HM, Shipley WU. Radiotherapy and short-term androgen deprivation for localized prostate cancer. N Engl J Med. 2011 Jul 14;365(2):107-18. doi: 10.1056/NEJMoa1012348. PMID 21751904
- [Result] McGowan D, Hunt D, Jones C, et al.: Effect of short-term endocrine therapy prior to and during radiation therapy on overall survival in patients with T1b-T2b adenocarcinoma of the prostate and PSA equal to or less than 20: initial results of RTOG 94-08. [Abstract] 2010 Genitourinary Cancers Symposium, March 5-7, 2010, San Francisco, California. A-6, 2010.
- [Derived] Spratt DE, Tang S, Sun Y, Huang HC, Chen E, Mohamad O, Armstrong AJ, Tward JD, Nguyen PL, Lang JM, Zhang J, Mitani A, Simko JP, DeVries S, van der Wal D, Pinckaers H, Monson JM, Campbell HA, Wallace J, Ferguson MJ, Bahary JP, Schaeffer EM, Sandler HM, Tran PT, Rodgers JP, Esteva A, Yamashita R, Feng FY. Artificial Intelligence Predictive Model for Hormone Therapy Use in Prostate Cancer. NEJM Evid. 2023 Aug;2(8):EVIDoa2300023. doi: 10.1056/EVIDoa2300023. Epub 2023 Jun 29. PMID 38320143
- [Derived] Jones CU, Pugh SL, Sandler HM, Chetner MP, Amin MB, Bruner DW, Zietman AL, Den RB, Leibenhaut MH, Longo JM, Bahary JP, Rosenthal SA, Souhami L, Michalski JM, Hartford AC, Amin PP, Roach M 3rd, Yee D, Efstathiou JA, Rodgers JP, Feng FY, Shipley WU. Adding Short-Term Androgen Deprivation Therapy to Radiation Therapy in Men With Localized Prostate Cancer: Long-Term Update of the NRG/RTOG 9408 Randomized Clinical Trial. Int J Radiat Oncol Biol Phys. 2022 Feb 1;112(2):294-303. doi: 10.1016/j.ijrobp.2021.08.031. Epub 2021 Sep 1. PMID 34481017

RESULTS

PARTICIPANT FLOW:
Groups:
- Hormone Therapy + Radiation Therapy: Neoadjuvant total androgen suppression (TAS) - Flutamide and Zoladex or Lupron - two months before and during radiation therapy.
Period: Overall Study
Arm/Group | Hormone Therapy + Radiation Therapy | Radiation Therapy Alone
Started | 1013 | 1015
Completed | 987 (Subjects with data available for the primary analysis are considered to have completed the study.) | 992 (Subjects with data available for the primary analysis are considered to have completed the study.)
Not Completed | 26 | 23
Not completed — Protocol Violation | 19 | 17
Not completed — Withdrawal by Subject | 7 | 6

BASELINE CHARACTERISTICS:
Population: All eligible patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Hormone Therapy + Radiation Therapy | Radiation Therapy Alone | Total
Number analyzed (Participants) | 987 | 992 | 1979
Age, Continuous [Median (Full Range); unit: years] | 70 [47 to 91] | 71 [47 to 88] | 71 [47 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 987 | 992 | 1979

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival Rate (10-year)
Description: Overall survival (OS) was calculated from randomization to the date of death from any cause and overall survival rates were estimated by the Kaplan-Meier method.
Time Frame: From date of randomization to 10 years
Population: All eligible patients.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Hormone Therapy + Radiation Therapy | Radiation Therapy Alone
Number analyzed (Participants) | 987 | 992
percentage of patients | 61.9 [58.3 to 65.3] | 56.8 [53.2 to 60.2]
Statistical Analysis 1: Comparison: Hormone Therapy + Radiation Therapy vs Radiation Therapy Alone; Null hypothesis: 8-year OS rate of 60% radiation therapy (RT) alone vs. 67% with hormone therapy. The study was designed with 90% power to detect a 7-percentage- point absolute difference in the 8-year survival rate, with the use of a one-sided log-rank test at the 0.025 significance level, requiring 1980 patients and 716 deaths for definitive analysis; Test type: Superiority; p = 0.0309, Log Rank; Hazard Ratio (HR) = 1.17, 95% CI 2-sided [1.01 to 1.35] — Reference level = Hormone Therapy + Radiation Therapy

2. Secondary Outcome: Disease-specific Survival Rate (10 Years)
Description: Disease-specific failure is defined as death certified as due to prostate cancer (by central review), death due to complications of treatment (irrespective of malignancy status), death from unknown causes with active malignancy, or death from unknown causes with previously documented relapse (either clinical or biochemical). Survival rates were estimated by means of cumulative incidence functions.
Time Frame: From registration to 10 years
Population: All eligible patients.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Hormone Therapy + Radiation Therapy | Radiation Therapy Alone
Number analyzed (Participants) | 987 | 992
percentage of participants | 95.7 [94.3 to 97.2] | 92.6 [90.8 to 94.4]
Statistical Analysis 1: Comparison: Hormone Therapy + Radiation Therapy vs Radiation Therapy Alone; Gray's test was used to compare cumulative incidence between treatment arms (1-sided significance level of 0.025) and the Fine-Gray model was used to calculate hazard ratios; Test type: Superiority; p = 0.001, Gray's test; Hazard Ratio (HR) = 1.86, 95% CI 2-sided [1.27 to 2.74] — Reference level = Hormone Therapy + Radiation Therapy

3. Secondary Outcome: Local Progression Rate (10 Years)
Description: Local progression defined as documented local progression as determined by clinical exam . Failure rates were estimated by means of cumulative incidence functions.
Time Frame: From registration to 10 years
Population: All eligible patients.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Hormone Therapy + Radiation Therapy | Radiation Therapy Alone
Number analyzed (Participants) | 987 | 992
percentage of participants | 10.9 [8.8 to 12.9] | 16.1 [13.7 to 18.4]
Statistical Analysis 1: Comparison: Hormone Therapy + Radiation Therapy vs Radiation Therapy Alone; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0013, Gray's test; Hazard Ratio (HR) = 1.5, 95% CI 2-sided [1.17 to 1.93] — Reference level = Hormone Therapy + Radiation Therapy

4. Secondary Outcome: Distant Failure Rate (10 Years)
Description: Failure is defined as documented metastatic disease. Failure rates were estimated by means of cumulative incidence functions.
Time Frame: From registration to 10 years
Population: All eligible patients.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Hormone Therapy + Radiation Therapy | Radiation Therapy Alone
Number analyzed (Participants) | 987 | 992
percentage of participants | 5.5 [3.9 to 7.0] | 8.0 [6.2 to 9.8]
Statistical Analysis 1: Comparison: Hormone Therapy + Radiation Therapy vs Radiation Therapy Alone; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.035, Gray's test; Hazard Ratio (HR) = 1.45, 95% CI 2-sided [1.03 to 2.06] — Reference level = Hormone Therapy + Radiation Therapy

5. Secondary Outcome: Biochemical Failure Rate (10 Years)
Description: The Phoenix definition of biochemical failure was used - an increase in the prostate-specific antigen (PSA) level of >2 ng per milliliter above the nadir. Failure rates were estimated by means of cumulative incidence functions.
Time Frame: From registration to 10 years
Population: All eligible patients.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Hormone Therapy + Radiation Therapy | Radiation Therapy Alone
Number analyzed (Participants) | 987 | 992
percentage of participants | 26.3 [23.4 to 29.2] | 41.1 [37.9 to 44.4]
Statistical Analysis 1: Comparison: Hormone Therapy + Radiation Therapy vs Radiation Therapy Alone; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.001, Gray's test; Hazard Ratio (HR) = 1.74, 95% CI 2-sided [1.48 to 2.04] — Reference level = Hormone Therapy + Radiation Therapy

6. Secondary Outcome: Clinical Relapse Rate (10 Years)
Description: Clinical relapse is defined as local progression or distant metastases. Failure rates were estimated by means of cumulative incidence functions.
Time Frame: From registration to 10 years
Population: All eligible patients.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Hormone Therapy + Radiation Therapy | Radiation Therapy Alone
Number analyzed (Participants) | 987 | 992
percentage of participants | 15.0 [12.6 to 17.3] | 21.7 [19.1 to 24.4]
Statistical Analysis 1: Comparison: Hormone Therapy + Radiation Therapy vs Radiation Therapy Alone; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.001, Gray's test; Hazard Ratio (HR) = 1.5, 95% CI 2-sided [1.21 to 1.85] — Reference level = Hormone Therapy + Radiation Therapy

7. Secondary Outcome: Second Biochemical Relapse Rate (10 Years)
Description: Second biochemical relapse is as defined as follows (after initiation of salvage hormone therapy): A rise in PSA on at least two consecutive cases above the nadir (after initiation of salvage hormone therapy), with the rises in PSA exceeding 1 ng/ml above the nadir; or failure to reach 4 ng/L or less at 18 months. The rates of second biochemical relapse were estimated by means of cumulative incidence functions.
Time Frame: From registration to 10 years
Population: All eligible patients.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Hormone Therapy + Radiation Therapy | Radiation Therapy Alone
Number analyzed (Participants) | 987 | 992
percentage of participants | 2.7 [1.6 to 3.8] | 6.1 [4.4 to 7.7]
Statistical Analysis 1: Comparison: Hormone Therapy + Radiation Therapy vs Radiation Therapy Alone; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.001, Gray's test; Hazard Ratio (HR) = 2.06, 95% CI 2-sided [1.34 to 3.16] — Reference level = Hormone Therapy + Radiation Therapy

8. Secondary Outcome: Disease-free Survival Rate (10 Years)
Description: Disease-free failure is defined as documentation of progression (local progression, distant failure, and biochemical failure) or death from any cause. Disease-free survival rates were estimated by the Kaplan-Meier method.
Time Frame: From registration to 10 years
Population: All eligible patients.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Hormone Therapy + Radiation Therapy | Radiation Therapy Alone
Number analyzed (Participants) | 987 | 992
percentage of participants | 51.7 [48.1 to 55.1] | 39.5 [36.1 to 42.9]
Statistical Analysis 1: Comparison: Hormone Therapy + Radiation Therapy vs Radiation Therapy Alone; Treatment arms were compared using the log-rank test (one-sided significance level of 0.025); Test type: Superiority; p < 0.001, Log Rank; Hazard Ratio (HR) = 1.38, 95% CI 2-sided [1.22 to 1.56] — Reference level = Hormone Therapy + Radiation Therapy

9. Secondary Outcome: Positive Re-biopsy Rate at Two Years
Description: The rate of prostate rebiopsy at two years is defined as the proportion of patients whose results are positive among all eligible patients who had a repeat biopsy at two years. The rate was estimated separately in each arm.
Time Frame: From registration to two years
Population: All eligible patients who had a repeat biopsy at 2 years.
Measure: Number; unit: percentage of participants
Arm/Group | Hormone Therapy + Radiation Therapy | Radiation Therapy Alone
Number analyzed (Participants) | 439 | 404
percentage of participants | 20.2 | 38.9
Statistical Analysis 1: Comparison: Hormone Therapy + Radiation Therapy vs Radiation Therapy Alone; Test type: Superiority; p < 0.001, Chi-squared

ADVERSE EVENTS:
Description: Eligible patients who received treatment. Subjects experiencing more than one of a given adverse event are counted only once for that adverse event.
Groups:
- Neoadjuvant TAS 2 Months Before and During RT: Neoadjuvant Total Androgen Suppression (TAS) two months before and during radiation therapy
Arm/Group | Neoadjuvant TAS 2 Months Before and During RT | Radiation Therapy Alone
Serious Adverse Events (participants affected / at risk) | 33/1003 | 16/1003
Other Adverse Events (participants affected / at risk) | 975/1003 | 955/1003
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Neoadjuvant TAS 2 Months Before and During RT (N=1003) | Radiation Therapy Alone (N=1003)
Acute RT Toxicity: Hematologic: NOS (Blood and lymphatic system disorders) | 7 | 5
Hormone Toxicity: Hematologic : NOS (Blood and lymphatic system disorders) | 1 | 0
Late RT Toxicity: Hematologic: NOS (Blood and lymphatic system disorders) | 8 | 3
Acute RT Toxicity: Bowel: NOS (Gastrointestinal disorders) | 1 | 0
Late RT Toxicity: Bowel: NOS (Gastrointestinal disorders) | 1 | 3
Late RT Toxicity: Other GI: NOS (Gastrointestinal disorders) | 2 | 0
Late RT Toxicity: Other: NOS (General disorders) | 3 | 0
Hormone Toxicity: Liver : NOS (Hepatobiliary disorders) | 3 | 0
Acute RT Toxicity: Bladder: NOS (Renal and urinary disorders) | 4 | 4
Late RT Toxicity: Bladder: NOS (Renal and urinary disorders) | 12 | 0
Late RT Toxicity: Other GU: NOS (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Neoadjuvant TAS 2 Months Before and During RT (N=1003) | Radiation Therapy Alone (N=1003)
Acute RT Toxicity: Hematologic: NOS (Blood and lymphatic system disorders) | 127 | 67
Hormone Toxicity: Hematologic : NOS (Blood and lymphatic system disorders) | 172 | 0
Late RT Toxicity: Hematologic: NOS (Blood and lymphatic system disorders) | 135 | 109
Acute RT Toxicity: Bowel: NOS (Gastrointestinal disorders) | 439 | 501
Late RT Toxicity: Bowel: NOS (Gastrointestinal disorders) | 262 | 210
Acute RT Toxicity: Other: NOS (General disorders) | 135 | 138
Late RT Toxicity: Other: NOS (General disorders) | 84 | 99
Hormone Toxicity: Liver : NOS (Hepatobiliary disorders) | 93 | 0
Acute RT Toxicity: Bladder: NOS (Renal and urinary disorders) | 149 | 190
Late RT Toxicity: Bladder: NOS (Renal and urinary disorders) | 182 | 166
Hormone Toxicity: Impotence : NOS (Reproductive system and breast disorders) | 238 | 0
Late RT Toxicity: Other GU: NOS (Reproductive system and breast disorders) | 69 | 78
Hormone Toxicity: Hot flashes : NOS (Vascular disorders) | 295 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.